CLINICAL TRIAL: NCT04682249
Title: Systemic Chemotherapy Based on Oxaliplatin and 5-fluorouracil, Apatinib Plus Sintilimab for Metastasis ICC: a Single Arm Prospective Study
Brief Title: Systemic Chemotherapy, Apatinib Plus Sintilimab for Metastasis ICC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no patients enrolled
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shi Ming, Proffessor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SL077B
Record Dates: First submitted 2020-12-20; First posted 2020-12-23 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: ICC
Keywords: ICC; Systemic Chemotheray; Apatinib; Sintilimab
MeSH Terms: interventions — Neoadjuvant Therapy; sintilimab; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Systemic Chemotheray, Apatinib plus Sintilimab (Experimental)
  Interventions: Drug: Systemic Chemotherapy; Drug: Sintilimab; Drug: Apatinib

INTERVENTIONS:
Drug: Systemic Chemotherapy — Systemic Chemotherapy (Oxaliplatin#5-fluorouracil and leucovorin)
Drug: Sintilimab — Sintilimab
Drug: Apatinib — Apatinib

SUMMARY:
This study were designed to verify the better method of survival for metastatic ICC. Since the traditional method for metastatic ICC was GEMOX(first-line treatment from NCCN guideline), our previous study found similar results from FOLFOX (second-line treatment from NCCN guideline) compared with GEMOX.

Our current study were conducted for further investigation to verify the better method for metastatic ICC.

DETAILED DESCRIPTION:
ICC(Intrahepatic CholangioCarcinoma) patients with metastasis has a short survival time and poor prognosis after diagnosis. Treatment methods was few and far from satisfaction. The treatment recommended from NCCN guideline was GEMOX(Systemic Chemotheray) and clinical trials. Our previous study has demonstrate FOLFOX (Systemic Chemotheray based on Oxaliplatin#5- fluorouracil) has a similar survival and tumor response compared with GEMOX. Further study was needed to intensive confirmation of the result. We designed this study to demonstrate the hypothesis. Metastasis ICCs were recruited and screened by our criteria. All patients were treated with FOLFOX (Systemic Chemotheray based on Oxaliplatin#5-fluorouracil ), apatinib (one of tyrosine kinase inhibitors) plus sintilimab (one of PD-1 antibody).

Our study were designed to verify the better method of survival for metastatic ICC.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of ICC
* With distant metastasis
* Patients must have at least one tumor lesion that can be accurately measured according to mRECIST criteria.
* With no previous treatment
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* Not amendable to surgical resection ,local ablative therapy and any other cured treatment
* The following laboratory parameters:

Platelet count ≥ 60,000/μL Hemoglobin ≥ 8.5 g/dL Total bilirubin ≤ 30mmol/ L Serum albumin ≥ 32 g/L ASL and AST ≤ 6 x upper limit of normal Serum creatinine ≤ 1.5 x upper limit of normal INR ≤ 1.5 or PT/APTT within normal limits Absolute neutrophil count (ANC) >1,500/mm3

Exclusion Criteria:

* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of bleeding diathesis.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Objective response rate | 6 months

SECONDARY OUTCOMES:
Overall survival | 6 months
Progression-free survival | 6 months
Number of adverse events | 30 days
  Postoperative adverse events were graded based on CTCAE v4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center Sun Yat-sen University, Guangzhou, Guangdong, China